CLINICAL TRIAL: NCT02869308
Title: Determination of Left Ventricular Ejection Fraction Using Cardiac Angioscintigraphy: Comparison Between Measurements Obtained With Conventional Planar Scintigraphy (E-CAM Camera) and Tomoscintigraphy Recorded by a CZT Semiconductor Camera (D-SPECT)
Brief Title: Determination of Left Ventricular Ejection Fraction Using Cardiac Angioscintigraphy
Acronym: FEVED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00650-45
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Angioscintigraphy; Tomoscintigraphy
Keywords: Cardiomyopathy; Chemotherapy; Left ventricular ejection fraction
MeSH Terms: conditions — Cardiomyopathies | interventions — Tin Polyphosphates; Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocardial angioscintigraphy (Other)
  Interventions: Drug: stannous pyrophosphate; Drug: Technetium-99m; Device: E-CAM Camera; Device: CZT Semiconductor Camera (D-SPECT)

INTERVENTIONS:
Drug: stannous pyrophosphate — Injection of 1ml Angiocis
  Other Names: Angiocis
Drug: Technetium-99m — Injection of 900 MBq Technetium-99m, 30 min after Angiocis injection
Device: E-CAM Camera — Acquisition of images of angioscintigraphy with E-CAM camera, after injection of Angiocis and Technetium-99m
Device: CZT Semiconductor Camera (D-SPECT) — Acquisition of images of angioscintigraphy with D-SPECT camera

SUMMARY:
The purpose is to determine whether measurements of left ventricular ejection fraction (LVEF) obtained with angiographies recorded by conventional Anger camera or D-SPECT camera are equivalent.

Secondary purposes are:

* To evaluate the influence of cardiac activity recorded by D-SPECT camera on equivalences defined in primary purpose
* To evaluate the influence of the indication for the examination with a distinct analysis of a group having the examination for a known or suspected cardiomyopathy (LVEF often abnormally low) and a group having the examination for a chemotherapy supervision with heart initially considered healthy (LVEF often normal).

DETAILED DESCRIPTION:
Cardiac angioscintigraphy is an examination for a simple, precise and reproducible measurement of left ventricular ejection fraction (LVEF). It needs injection of 99mTc labeled albumin or red cells and unfortunately injected activities must be relatively considerable (≈ 900 MBq) for image recording times shorter than 10 minutes. This examination is thus quite irradiant (10 mSv) but this inconvenient could be eliminated with new semiconductor cameras.

These new cameras allow a better image quality than conventional Anger cameras (better spatial resolution and energy) and their detection sensitivity is almost 10 times higher. However, these new cameras can record only 3D images whereas with conventional cameras angioscintigraphy is usually performed in bidimensional way with a possible higher precision and reproducibility of LVEF measurement.

In this study, patients needing the routine examination for LVEF measurements will undergo the conventional examination followed by examination with semiconductor camera (without supplementary injection).

If LVEF measurement with semiconductor camera will be as precise and reproducible as with conventional camera, angioscintigraphy could be performed with these new cameras with a lower body irradiation of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients present in Nuclear Medicine department for measurement of LVEF by cardiac angioscintigraphy for known or suspected cardiomyopathy or for a chemotherapy supervision with heart initially considered healthy
* Without guardianship, signed informed consent
* Not in life-and-death emergency and with a stable clinical state
* Affiliated to social security
* Preliminary medical examination

Exclusion Criteria:

* Patients having rhythm disorders (atrial or ventricular extrasystoles in more than 20% cardiac cycles, atrial fibrillation)
* Incapable to stay in strict decubitus position during image recording times
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of measurement of LVEF with conventional camera and semiconductor camera analyzed by two different person | day 0

SECONDARY OUTCOMES:
Measurements of LVEF with cardiac activity recorded by D-SPECT camera artificially diminished of 25% | day 0
Measurements of LVEF with cardiac activity recorded by D-SPECT camera artificially diminished of 50% | day 0
Measurements of LVEF with cardiac activity recorded by D-SPECT camera artificially diminished of 75% | day 0
Comparison of measurements of LVEF with conventional camera and semiconductor camera in group of patients having cardiomyopathies | day 0
Comparison of measurements of LVEF with conventional camera and semiconductor camera in group of patients under LVEF supervision for chemotherapy | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Gilles KARCHER, Pr, Principal Investigator — CHU de NANCY - Service de Médecine Nucléaire - France
Locations (1):
- CHU de NANCY - Service de Médecine Nucléaire, Nancy, France

IPD SHARING:
Plan to Share IPD: No